CLINICAL TRIAL: NCT02008825
Title: Evaluation of the ViSiGiTM Calibration System for Effectiveness With Sleeve Visual Delineation at Various Suction Levels.
Brief Title: Evaluation of the ViSiGiTM Calibration System
Acronym: ViSiGi
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Luke's Hospital and Health Network, Pennsylvania (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Leonardo Claros, Bariatric Section Chief and Program Director, St. Luke's Hospital and Health Network, Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLHN2013-62
Record Dates: First submitted 2013-11-07; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Enhance Delineation of the Stomach Anatomy and the Surgeon's Appreciation of the Extent of Gastric Volume to be Removed;; Increase the Safety Profile of the Patient (i.e., Reduce the Likelihood of Accidental Stapling of the Orogastric Tube or Bougie);; Reduce the Incidence of OR Contamination/Infection Transmission;; Streamline OR Workflow, Resulting in Reduced OR Time; Ensure Consistent and Reproducible Staple Lines.
Keywords: ViSiGi; Calibration tube; Sleeve gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ViSiGi (Experimental): Utilization of ViSiGi calibration tube
  Interventions: Device: Utilization of ViSiGi calibration tube
- Usual standard of care (Active Comparator): Usual non suction Bougie
  Interventions: Device: Usual non suction Bougie

INTERVENTIONS:
Device: Utilization of ViSiGi calibration tube — Utilization of ViSiGi calibration tube
  Other Names: ViSiGi 3D
  Arms: ViSiGi
Device: Usual non suction Bougie — Usual non suction Bougie
  Arms: Usual standard of care

SUMMARY:
We hypothesize that using the ViSiGi™ Calibration Tube System in patients undergoing LSG will:

1. enhance delineation of the stomach anatomy and the surgeon's appreciation of the extent of gastric volume to be removed;
2. increase the safety profile of the patient (i.e., reduce the likelihood of accidental stapling of the orogastric tube or bougie);
3. reduce the incidence of OR contamination/infection transmission;
4. streamline OR workflow, resulting in reduced OR time; and
5. ensure consistent and reproducible staple lines.

DETAILED DESCRIPTION:
Laparoscopic Sleeve Gastrectomy (LSG), is now widely used as a stand-alone procedure for long-term weight loss. With fewer potential morbidities, comparable weight loss and greater ease of conversion to other procedures, many patients now opt for LSG as their bariatric procedure of choice. During surgery gastric decompression and calibration are compulsory for patient safety, gastric anatomic delineation, ease of surgery and optimal weight loss. The removed gastric volume at surgery seems to predict the procedure's success rates2. LSG performed without calibration (tube) could result in inconsistent staple lines, with retained high sleeve volume and consequent failure. Traditionally, although different tubes are used for gastric decompression and calibration, this protocol interrupts operation room (0R) workflow. Accidental stapling of orogastric tubes and bougies do occur in the OR but are seldom reported. The need for this multiple tube system can be obviated with the ViSiGi™ Calibration Tube System. A single, multipurpose tube that integrates all these various steps could prevent breaks in OR; improve workflow; reduce patient injuries, cross contamination and transmission of infections; and a consistent and reproducible staple line. A similar device has been in use in Europe, Australia and Asia, but the ViSiGi™ Calibration Tube System is the first of its kind to be approved by the FDA. Currently, there are no data on its clinical safety/efficacy in comparison to standard care of separate orogastric tube and bougie in the United States. Therefore, this exploratory study will investigate the gastric delineation ability, general safety and efficacy of the ViSiGi™ Calibration Tube System along with the regular bougie in LSG patients over a six- to twelve-month period. Descriptive outcomes will be reported, with no formal sample size calculation in light of the exploratory study design.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide written informed consent for study participation.
* age 18 years or older
* candidate for laparosopic gastrectomy with no history of previous bariatric surgeries (i.e., gastric bypass, band, duodenal switch)attendance at an informational seminar and support group
* clearance for surgery by a registered dietician and certified social worker
* BMI > 35 with at least one co-morbid condition (e.g., hypertension, diabetes mellitus, sleep apnea, hypercholesterolemia) or BMI > 40 without any co-morbid conditions
* negative pregnancy test
* American Society of Anesthesiology score 1-3
* ability to understand instructions and comply with all study requirements
* pre-operative %excess weight loss (%EWL) of 3-10%
* no contraindication for LSG based on upper endoscopy findings
* pre-operative cardiac consultation for risk stratification
* evaluation by a sleep medicine specialist to identify risk factors for sleep apnea, with treatment as deemed appropriate

Exclusion Criteria:

* current participation in another clinical trial that involves any investigational drug or device that would interfere with this study
* Barrett's Esophagus, severe gastric paresis/atony, achalasia, neoplasm or other complications discovered during preoperative esophago-gastro-duodonoscopy.
* revisional surgery
* conversion to open procedure
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Efficasy | 3 months
  This exploratory study will investigate the gastric delineation ability, general safety and efficacy of the ViSiGi™ Calibration Tube System along with the regular bougie in LSG patients over a six- to twelve-month period. Descriptive outcomes will be reported, with no formal sample size calculation in light of the exploratory study design.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luke's University and Health Network, Allentown, Pennsylvania, United States

REFERENCES:
- [Background] Satiani B, Bonner JT, Stone HH. Factors influencing intraoperative gastric regurgitation: a prospective random study of nasogastric tube drainage. Arch Surg. 1978 Jun;113(6):721-3. doi: 10.1001/archsurg.1978.01370180063008. PMID 26318
- [Background] Weiner RA, Weiner S, Pomhoff I, Jacobi C, Makarewicz W, Weigand G. Laparoscopic sleeve gastrectomy--influence of sleeve size and resected gastric volume. Obes Surg. 2007 Oct;17(10):1297-305. doi: 10.1007/s11695-007-9232-x. PMID 18098398
- [Background] Abu-Gazala S, Donchin Y, Keidar A. Nasogastric tube, temperature probe, and bougie stapling during bariatric surgery: a multicenter survey. Surg Obes Relat Dis. 2012 Sep-Oct;8(5):595-600; discussion 600-1. doi: 10.1016/j.soard.2011.08.017. Epub 2011 Aug 31. PMID 21963196
- [Background] Pequignot A, Dhahria A, Mensah E, Verhaeghe P, Badaoui R, Sabbagh C, Regimbeau JM. Stapling and Section of the Nasogastric Tube during Sleeve Gastrectomy: How to Prevent and Recover? Case Rep Gastroenterol. 2011;5(2):350-4. doi: 10.1159/000329706. Epub 2011 Jul 6. PMID 21769286
- [Background] Sanchez BS, Safadi BY, Kieran JA, Hsu GP, Brodsky JB, Curet MJ, Morton JM. Orogastric tube complications in laparoscopic Roux-en-Y gastric bypass. Obes Surg. 2006 Apr;16(4):443-7. doi: 10.1381/096089206776327350. PMID 16608608
- [Background] Vennes JA. Infectious complications of gastrointestinal endoscopy. Dig Dis Sci. 1981 Jul;26(7 Suppl):60S-64S. doi: 10.1007/BF01300809. PMID 6765053
- [Background] Kovaleva J, Peters FT, van der Mei HC, Degener JE. Transmission of infection by flexible gastrointestinal endoscopy and bronchoscopy. Clin Microbiol Rev. 2013 Apr;26(2):231-54. doi: 10.1128/CMR.00085-12. PMID 23554415
- [Background] Schembre DB. Infectious complications associated with gastrointestinal endoscopy. Gastrointest Endosc Clin N Am. 2000 Apr;10(2):215-32. PMID 10683209
- See also: ViSiGi web site — http://www.visigi.com